CLINICAL TRIAL: NCT07282483
Title: Traditional Chinese Medicine Oral Liquids and Mouthwashes for Radiation-induced Oral Mucositis in Head and Neck Cancer Patients: A Randomized Controlled Trial
Brief Title: Traditional Chinese Medicine Oral Liquids and Mouthwashes for Radiation-induced Oral Mucositis in Head and Neck Cancer Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, PhD, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-1774
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Radiation-induced Oral Mucositis
MeSH Terms: interventions — Mouthwashes; Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qingying oral liquid and modified Da Huang-Huang Lian Xiexin mouthwash (Active Comparator)
  Interventions: Drug: Qingying oral liquid and modified Da Huang-Huang Lian Xiexin mouthwash; Radiation: radiotherapy
- Placebo oral solution and mouthwash (Placebo Comparator)
  Interventions: Drug: Placebo oral solution and mouthwash; Radiation: radiotherapy

INTERVENTIONS:
Drug: Qingying oral liquid and modified Da Huang-Huang Lian Xiexin mouthwash — Classical traditional Chinese medicine (TCM) formulations provided as an oral liquid and a herbal mouthwash
  Arms: Qingying oral liquid and modified Da Huang-Huang Lian Xiexin mouthwash
Drug: Placebo oral solution and mouthwash — A placebo matched in color, odor, and taste to the Qingying oral liquid and the modified Da Huang-Huang Lian Xiexin mouthwash, but containing no active medicinal ingredients.
  Arms: Placebo oral solution and mouthwash
Radiation: radiotherapy — All subjects underwent radical radiotherapy

SUMMARY:
Evaluate the efficacy and safety of traditional Chinese medicine oral liquid and mouthwash in the treatment of radiotherapy induced oral mucositis in patients with head and neck malignancies

DETAILED DESCRIPTION:
The aim of this clinical trial is to evaluate the efficacy and safety of combining a traditional Chinese medicine (TCM) oral liquid with a mouthwash in reducing the incidence, duration, and severity of mild-to-moderate radiation-induced oral mucositis (RIOM). The study addresses two main questions: (1) whether the combined TCM oral liquid and mouthwash can effectively mitigate RIOM and lower the incidence of severe RIOM, and (2) whether their use is associated with adverse events in patients receiving radiotherapy.

Participants will begin treatment on the first day mild-to-moderate RIOM (RTOG grade 1-2) occurs during radiotherapy. They will take Qingying oral liquid four times daily and use a modified Da Huang-Huang Lian Xiexin mouthwash six times daily in combination, or receive a matching placebo. The treatment will continue until two weeks after radiotherapy. After each administration, patients must avoid eating, drinking, or performing oral hygiene for at least 1 hour to maximize mucosal contact time.

The trial will compare the intervention and placebo groups to determine the potential benefits of the combined regimen for managing RIOM.

ELIGIBILITY:
Inclusion Criteria:

1. Patients pathologically diagnosed with non-metastatic head and neck malignant tumors;
2. Age range: 18 to 65 years old (including 18 and 65 years old);
3. Eastern Cooperative Oncology Group performance status of ≤2;
4. Radiotherapy or concurrent chemoradiotherapy is required;
5. The main organ functions well;
6. Sign informed consent.

Exclusion Criteria:

1. Allergic constitution (such as those known to be allergic to two or more drugs);
2. Patients who plan to use drugs that can cause or worsen oral mucosal inflammation (such as anti EGFR monoclonal antibodies, immune checkpoint inhibitors, etc.) after the start of radiotherapy;
3. Use of antibiotics, antifungal drugs, or antimicrobial mouthwash within 1 month of the study;
4. Poor oral hygiene and/or severe periodontal diseases;
5. History of head and neck radiotherapy;
6. Deemed unsuitable for the study by the investigators (concomitant with any other severe diseases).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of severe oral mucositis (RTOG grade ≥ 3) | From the start of radiotherapy to 8 weeks after the end of radiotherapy. The evaluation period is approximately 14 to 14.5 weeks
  The Radiation Therapy Oncology Group (RTOG) toxicity criteria were utilized to assess RIOM. Grade 0 shows no change from baseline; Grade 1 of RIOM is associated with mucosal erythema or hyperemiam,and may cause mild pain not requiring analgesics. Grade 2 presents with patchy mucositis that may produce an inflammatory serosanguinous discharge and may be associated with moderate pain; Grade 3 consists of confluent, fibrinous mucositis and may include severe pain requiring narcotics; Grade 4 is characterized by ulceration, hemorrhage, or necrosis. Grades 1 and 2 are considered mild to moderate, while grades 3 and 4 are classified as severe.

SECONDARY OUTCOMES:
Duration of mild-to-moderate RIOM | From the start of radiotherapy to 8 weeks after the end of radiotherapy. The evaluation period is approximately 14 weeks and 14.5 weeks.
  Time from the first documentation of RTOG grade 1-2 oral mucositis during radiotherapy to the first return to RTOG grade 0 (no mucositis) sustained for ≥48 hours.
RIOM remission rates at 4 and 8 weeks after completion of radiotherapy | From the start of radiotherapy to 8 weeks after the end of radiotherapy. The evaluation period is approximately 14 weeks and 14.5 weeks.
  The proportion of participants whose oral mucositis has decreased to RTOG grade 0 at 4 and 8 weeks after completion of radiotherapy, respectively.
Duration of oral mucositis (OM) | From the start of radiotherapy to 8 weeks after completion of radiotherapy.The evaluation period is approximately 14 weeks and 14.5 weeks.
  The first determination of OM to the first instance of non-OM, without a subsequent instance of OM.
Weekly change in oropharyngeal pain scores (OMWQ) | From the start of radiotherapy to 8 weeks after completion of radiotherapy.The evaluation period is approximately 14 weeks and 14.5 weeks.
  Patients report mouth and throat soreness (MTS) scores (Likert scale 1 to 5) via the oral mucositis weekly questionnaire （OMWQ）. Higher score indicates more severe symptoms
Use of analgesics | From the start of radiotherapy to 8 weeks after completion of radiotherapy.The evaluation period is approximately 14 weeks and 14.5 weeks.
  Recorded as any use (yes/no), agent class, daily dose standardized to oral morphine milligram equivalents (MME), and total days of use during radiotherapy and through 8 weeks post-radiotherapy.
Xerostomia | 1 week before radiotherapy ; at the middle of radiotherapy (3 weeks after the start of radiotherapy) ; at the end of radiotherapy (the last radiation dose received, usually 6 or 6.5 weeks); 4 weeks and 8 weeks after the end of radiotherapy.
  Xerostomia was graded per CTCAE v5.0 (Grade 1-4), with higher grades indicating worse symptoms.
European Organization for Research and Treatment of Cancer (EORTC) Head and Neck Cancer Module (EORTC QLQ-H&N35). | 1 week before radiotherapy ; at the middle of radiotherapy (3 weeks after the start of radiotherapy) ; at the end of radiotherapy(the last radiation dose received, usually 6 or 6.5 weeks) ; and and 4 weeks and 8 weeks after the end of radiotherapy.
  Quality of life questionnaire
Adverse events | From the first day of radiotherapy to the day of the last radiation dose received, usually 6 or 6.5 weeks.
  Common Terminology Criteria for Adverse Events (CTCAE) 5.0 version

OTHER OUTCOMES:
The longitudinal dynamics of salivary microbiota | 1 week before radiotherapy, the middle of radiotherapy (3 weeks after the start of radiotherapy), and the end of radiotherapy (the last radiation dose received, usually 6 or 6.5 weeks).
  Unstimulated whole saliva samples will be collected via spitting method at three time points: baseline, mid-term radiotherapy (the week corresponding to 50% completion of the planned radiation fractions), and the end of radiotherapy (the final week of RT). 16S rRNA gene sequencing will be performed to assess alterations in the oral microbiota.
TCM syndrome score for RIOM | From the start of radiotherapy to 8 weeks after completion of radiotherapy.The evaluation period is approximately 14 weeks and 14.5 weeks.
  Analyze patients' post-radiotherapy TCM syndromes using the Radiation-Induced Oral Mucositis Syndrome Scale.
Analysis of Inflammatory Indicators in Oral Saliva | 1 week before radiotherapy, the middle of radiotherapy (3 weeks after the start of radiotherapy), and the end of radiotherapy (the last radiation dose received, usually 6 or 6.5 weeks).
  Measurement of circulating levels of interleukin-1β (IL-1β), interleukin-6 (IL-6), and tumor necrosis factor-alpha (TNF-α) in patient oral saliva.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuan, China